CLINICAL TRIAL: NCT00101530
Title: Partnership Programs to Reduce Cardiovascular Disparities - Latinos Using Cardio Health Actions to Reduce Risk
Brief Title: Improving Prevention of Heart Disease in Latinos
Acronym: LUCHAR
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-0621; U01HL079208 (NIH); U01HL079160 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to improve cardiovascular disease (CVD) outcomes in racial and ethnic minorities. Specifically, it seeks to improve the primary prevention of CVD in Hispanics.

DETAILED DESCRIPTION:
BACKGROUND:

While there has been great progress in reducing CVD morbidity and mortality in the United States over the past 40 years, some minority groups have not shared fully in this progress and continue to have lower life expectancy and higher CVD morbidity. On average, minorities have less access to medical care, receive less aggressive care and fewer diagnostic and therapeutic cardiac procedures, and adhere poorly to prescribed medical regimens. Thus, research to reduce health disparities by improving CVD outcomes in minorities offers potential for a substantial positive public heath impact. Academic medical centers and institutions capable of carrying out such research, however, often lack access to and the trust of minority patients. Minority patients often receive fragmented care because they lack access to regular medical care, present to emergency departments rather than primary care physicians for complications of an advanced chronic CVD condition, and are less likely to follow medical regimens. Minority communities often harbor distrust of clinical research. Minority patients report greater satisfaction when receiving care from minority providers and are reluctant to receive treatment outside their minority health care serving systems.

In general, minorities have high rates of hypertension, elevated cholesterol, cigarette smoking, obesity, metabolic syndrome, and diabetes as well as other behavioral, environmental, and occupational risk factors for cardiovascular diseases, such as sleep problems - all elements that contribute to excess CVD morbidity and mortality. The causes of minority health disparities are complex and incompletely understood. Although evidence of genetic, biologic, and environmental factors is well documented, poor outcomes are also attributed to undertreatment. Such undertreatment may be due to limited access to health care or, in some cases, breakdown of the medical system, or failure of the physician and/or patient to allow for optimal health care, even when access is not impaired. The complex interactions of behavior, socioeconomic status (SES), culture, and ethnicity are important predictors of health outcomes and sources of health disparities. Despite efforts to elucidate genetic and environmental risk factors and to promote cardiovascular health in high-risk populations, trends in CVD outcomes suggest that CVD health disparities continue to widen.

The Partnerships Program to Reduce Cardiovascular Health Disparities involves collaboration between research-intensive medical centers (RIMCs) that have a record of NIH-supported research and patient care and minority health care serving systems (MSSs) that lack a strong research program. Each Partnership Program will (a) design and carry out multiple interdisciplinary research projects that investigate complex biological, behavioral, and societal factors that contribute to CVD health disparities and facilitate clinical research within the MSS to improve CVD outcomes and reduce health disparities and (b) provide reciprocal educational and skills development programs so that investigators are able to conduct research aimed at reducing cardiovascular disparities and thereby enhance research opportunities and enrich cultural sensitivity and cardiovascular research capabilities at both institutions.

The Request for Applications for Partnership Programs to Reduce Cardiovascular Disparities was released in September 2003. The awards were made in September 2004.

DESIGN NARRATIVE:

The study will develop a partnership between Denver Health (DH), an MSS, and the University of Colorado Health Sciences Center (UCHSC), an RIMC. The first specific aim of the project is to develop and evaluate an interactive computer-based tool to improve community-based recognition of cardiovascular risk factors and to improve self-management skills, including adherence with clinic visits. The tool will be culturally sensitive and bilingual. The second specific aim is to test the ability of a nurse-based disease management program to improve control of risk factors. Under this aim, DH's unique computerized information system will be used to develop a registry of patients with hypertension and to characterize patients' overall risk for CVD and their risk for nonadherent behavior. A randomized clinical trial will be used to assess the impact of a nurse-based disease management intervention in those at highest risk and with a history of nonadherence. The intervention will be based on programs already in place at DH but will be modified in response to input from community-based focus groups. Specific aims 3 and 4 will seek to refine current cardiovascular risk profiling in ways specific to Hispanics. Specific aim 3 will assess ethnic differences in the relationship between traditional risk factors (diabetes, hypertension, smoking, and hyperlipidemia) and preclinical markers of cardiovascular disease (left ventricular mass, carotid intima media thickness, and brachial artery reactivity) over time. Specific aim 4 will assess the relationship among the traditional risk factors, preclinical markers, and a panel of circulating inflammatory markers. Also under specific aim 4, a randomized, placebo-controlled trial will assess the efficacy of "statin" medications to reduce circulating levels of these inflammatory markers. Specific aims 5 and 6 will develop educational programs to increase the cultural proficiency of clinical researchers, increase minority researcher participation in cardiovascular prevention research, and assist junior DH physicians in developing research careers in cardiovascular prevention.

ELIGIBILITY:
Eligibility Criteria vary with each study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: White and Latino patients in a safety net hospital
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2004-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Havranek, MD, Principal Investigator — Denver Health and Hospital Authority; Sheana Bull, PhD, Principal Investigator — University of Colorado Denver/HSC Aurora
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States